CLINICAL TRIAL: NCT05060354
Title: Immune Response to SARS-CoV2 Vaccinations in Treated MS Patients Compared to Controls
Brief Title: COVID-19 Vaccine Response in Treated MS Patients
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tanuja Chitnis, Senior Neurologist, Professor of Neurology, Brigham and Women's Hospital
Other Study IDs: COMB157GUS19T
Record Dates: First submitted 2021-09-27; First posted 2021-09-29 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis; Healthy
Keywords: Multiple Sclerosis; COVID-19; mRNA vaccine
MeSH Terms: conditions — Multiple Sclerosis; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Approximately 120 mL whole blood will be collected from each subject at each timepoint: 20 mL will be sent to the BWH clinical laboratories for same day SARS-CoV2 antibody assays and immunoglobulin levels. Additional blood for research immune assays will be collected and stored: 60-70 mL will be collected in cell preparation tubes (CPTs) for peripheral blood mononuclear cell (PBMC) isolation, 10 mL for DNA isolation and 20 mL by serum separator tubes for serum collection using a standardized sample collection kit. PBMCs will isolated and stored in liquid nitrogen and serum will be frozen at -80 °C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MS Kesimpta (ofatumumab): MS patients treated with Kesimpta (ofatumumab) for at least 3 months prior to SARS-CoV2 vaccination (completed regimen) Drug administration n/a, following routine clinical care Blood draws at 2-3 months, 5-6 months, and 11-12 months after enrollment
  Interventions: Other: Blood draw
- MS Ocrevus (ocrelizumab): MS patients treated with Ocrevus (ocrelizumab) for at least 3 months prior to SARS-CoV2 vaccination (completed regimen) Drug administration n/a, following routine clinical care Blood draws at 2-3 months, 5-6 months, and 11-12 months after enrollment
  Interventions: Other: Blood draw
- MS Gilenya (fingolimod) and Mayzent (siponimod): MS patients treated with Gilenya (fingolimod) or Mayzent (siponimod) for at least 3 months prior to SARS-CoV2 vaccination (completed regimen) Drug administration n/a, following routine clinical care Blood draws at 2-3 months, 5-6 months, and 11-12 months after enrollment
  Interventions: Other: Blood draw
- Healthy Control: Individuals with major autoimmune disorders or current treatment with immunosuppressive or immunomodulatory drugs Received SARS-CoV2 vaccination (completed regimen) within 2-6 months of enrollment Blood draws at 2-3 months, 5-6 months, and 11-12 months after enrollment
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Approximately 120 mL whole blood will be collected from each subject at each timepoint

SUMMARY:
The primary goal of this study is to assess the impact of the two major disease modifying therapy (DMT) classes (B cell therapies and S1P modulators) on humoral and cell-mediated immunity to SARS- CoV-2 vaccination compared to non-MS controls. We have chosen to compare DMT-treated MS patients to non-MS controls because the pivotal vaccine studies were conducted in non-MS healthy control groups in which there is significant clinical data and validated assays for antibody responses.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) affects approximately 1 million persons in the United States and is the leading cause of disability in young adults. Disease modifying treatments for MS act through modulation or suppression of immune responses including B and T cell responses. Two major classes of drugs used to treat MS are 1) B cell antibodies, including Kesimpta (ofatumumab) and Ocrevus (ocrelizumab), and 2) S1P (sphingosine-1-phosphate) modulators including Gilenya (fingolimod) and Mayzent (siponimod). SARS-CoV2 is a potentially fatal novel coronavirus, which has claimed over 350,000 lives in the United States. The causative agent of COVID-19 disease, the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) utilizes the angiotensin converting enzyme II (ACE2) to target cells in the lower airway.(1, 2) Symptoms of COVID-19 infection can cause pneumonia with primarily lymphocytic inflammatory infiltrates.(3) Most people (approximately 81%) experience mild upper respiratory tract infection or mild pneumonia, while approximately 15-20% of cases experience severe or critical disease characterized by dyspnea, lung infiltrates, respiratory failure and multiple organ dysfunction.(4) The case- fatality rate ranges from 0.7-5.8%. SARS-CoV2 vaccines have just been FDA approved, including the Moderna® and Pfizer-BioNTech® vaccines which contain lipid nanoparticle- formulated nucleoside-modified mRNA (messenger ribonucleic acid) that encodes the receptor binding domain (RBD) of the SARS-CoV-2 spike protein.(5, 6) Prior work suggests that vaccine responses may be blunted in patients treated with these two drug classes, however there is currently no controlled data on the efficacy and durability of SARS-CoV2 vaccine responses in treated MS patients. Current data is limited to uncontrolled case reports.

Robust studies are needed to inform the efficacy of SARS-CoV2 vaccines in MS patients on DMTs, which will guide infection risk management.

The primary goal of this study is to assess the impact of the two major DMT classes (B cell therapies and S1P modulators) on humoral and cell-mediated immunity to SARS- CoV-2 vaccination compared to non-MS controls. We have chosen to compare DMT-treated MS patients to non-MS controls because the pivotal vaccine studies were conducted in non-MS healthy control groups in which there is significant clinical data and validated assays for antibody responses.

The primary endpoint of this study is to compare the percentage of MS patients on immunotherapy with a positive SARS-CoV-2 Spike antibody response (positive seroconversion) compared to the percentage of controls who seroconvert at 5-6 months post vaccination.

Secondary endpoints of this study are:

* Comparison of SARS-CoV-2 Spike antibody % seroconversion and titers in MS patients on immunotherapy to titers in controls at 2-3 months and 11-12 months post vaccination.
* Comparison of T cell responses to SARS-CoV-2 spike protein in MS patients on immunotherapy to titers in controls at 5-6 months post vaccination.
* Comparison of antibody titers and T cell responses between the four groups of immunotherapies evaluated and to controls at each of the three timepoints.

ELIGIBILITY:
Inclusion Criteria:

For MS Patients:

1. Diagnosis of MS
2. Treatment with one of the four DMTs (Kesimpta (ofatumumab), Ocrevus (ocrelizumab), Gilenya (fingolimod), Mayzent (siponimod)) for at least 3 months prior to first SARS-CoV2 vaccine dose
3. SARS-CoV2 vaccine regimen complete within the past 2-3 or 5-6 months (either Moderna® or Pfizer-BioNTech® mRNA vaccines)
4. Age 18-65, inclusive

For Health Controls:

1. Age 18-65, inclusive

Exclusion Criteria:

For MS Patients:

1. Prior known COVID-19 infection

For Health Controls:

1. Prior known COVID-19 infection
2. major autoimmune disorders or current treatment with immunosuppressive or immunomodulatory drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For this study, we will prospectively collect data and biospecimens from MS patients and healthy volunteers. MS patients will largely be recruited from the Brigham MS Center at Brigham and Women's Hospital (Boston MA US). Healthy volunteers will be recruited from the community surrounding BWH and through IRB-approved recruitment advertisements. The Brigham MS Center sees 2500 patients annually and is adjacent to an ongoing COVID vaccine clinic.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Primary endpoint | 11-12 months
  Compare the percentage of MS patients on immunotherapy with a positive SARS-CoV-2 Spike antibody response, using the Roche Elecsys® Anti-SARS-CoV-2 S immunoassay for the quantitative, in vitro determination of antibodies to SARS-CoV- 2 in human serum and plasma. It is an Electro-chemiluminescence immunoassay (ECLIA) test using a double-antigen sandwich assay. A positive seroconversion defined as level>0.4U/ml.

SECONDARY OUTCOMES:
Secondary endpoint 1 | 11-12 months
  Comparison of SARS-CoV-2 Spike antibody % seroconversion and titers in MS patients on immunotherapy to titers in controls at 2-3 months and 11-12 months post vaccination. This will be measured as a percentage.
Secondary endpoint 2 | 5-6 months
  Comparison of percentage of IFN-gamma positive CD4+ T cells measured by flow cytometry reactive to SARS-CoV-2 spike protein in MS patients on immunotherapy to titers in controls at 5-6 months post vaccination.
Secondary endpoint 3 | 11-12 months
  Comparison of antibody titers and percentage of IFN-gamma positive CD4+ T cells reactive to SARS-CoV-2 measured by flow cytometry between the four groups of immunotherapies evaluated and to controls at each of the three timepoints 2-3, 5-6, and 11-12 months.
Secondary endpoint 4 | 11-12 months
  Comparison of SARS-CoV-2 Spike antibody seroconversion and levels in MS patients on immunotherapy after 2 vaccine doses versus 3 or more vaccine doses, as measured by Roche Elecsys® Anti-SARS-CoV-2 S immunoassay, with a positive seroconversion defined as >0.4U/ml.
Secondary endpoint 5 | 11-12 months
  Comparison of percentage SARS-CoV-2 reactive IFN-gamma positive CD4+ T cells measured by flow cytometry in MS patients on immunotherapy after 2 vaccine doses versus 3 or more vaccine doses.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham MS Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Derived] Conway S, Saxena S, Baecher-Allan C, Krishnan R, Houtchens M, Glanz B, Saraceno TJ, Polgar-Turcsanyi M, Bose G, Bakshi R, Bhattacharyya S, Galetta K, Kaplan T, Severson C, Singhal T, Stazzone L, Zurawski J, Paul A, Weiner HL, Healy BC, Chitnis T. Preserved T cell but attenuated antibody response in MS patients on fingolimod and ocrelizumab following 2nd and 3rd SARS-CoV-2 mRNA vaccine. Mult Scler J Exp Transl Clin. 2023 Apr 5;9(2):20552173231165196. doi: 10.1177/20552173231165196. eCollection 2023 Apr-Jun. PMID 37057191
- See also: Network recruitment site — https://rally.partners.org/study/covid